CLINICAL TRIAL: NCT02003235
Title: Assessment of Device for Treatment of Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visior Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-TMSC-1
Record Dates: First submitted 2013-12-01; First posted 2013-12-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Amblyopia
Keywords: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Daily watching videos using Reviview™, a dichoptic video display device
  Interventions: Device: Daily watching videos using Reviview™, a dichoptic video display device, for 60 min

INTERVENTIONS:
Device: Daily watching videos using Reviview™, a dichoptic video display device, for 60 min

SUMMARY:
The study will evaluate the effect of Reviview™, a dichoptic video display device for administrating a novel treatment protocol for Amblyopia (lazy eye) in kids.

The effect of the treatment will be measured by the change from baseline in Visual acuity and in Stereoscopic Vision; and to assess the ease of use of and compliance by the patients.

ELIGIBILITY:
Inclusion Criteria:

Refractive or Strabismic Amblyopia, with best corrected visual acuity.

(1) Refractive Amblyopia, visual acuity score <6:15 (worse then)

* or (2) Strabismic Amblyopia, visual acuity score between 6:15 and 6:30

Exclusion Criteria:

Diagnosed with epilepsy, recently treated with occlusion or penalization therapy

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Improvement in VA in amblyopic eye | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Haim Stolovitch, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel